CLINICAL TRIAL: NCT00129519
Title: Open-label Study to Evaluate the Use of Imiquimod 5% Cream for Reducing Postsurgical Recurrence or Persistence of Basal Cell Carcinoma Following Excision by Curettage
Brief Title: A Study to Evaluate the Effectiveness of Imiquimod 5% Cream for Basal Cell Carcinoma Recurrence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Graceway Pharmaceuticals, LLC (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1491-IMIQ
Record Dates: First submitted 2005-08-11; First posted 2005-08-12 (Estimated); Last update posted 2010-07-16 (Estimated); Status verified 2010-07

CONDITIONS: Basal Cell Carcinoma
Keywords: BCC curettage
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imiquimod cream (Active Comparator): Imiquimod 5% cream applied once daily 5x/week for up to 6 weeks
  Interventions: Drug: Imiquimod 5% cream

INTERVENTIONS:
Drug: Imiquimod 5% cream — Imiquimod 5% cream applied once daily 5x/week for up to 6 weeks

SUMMARY:
The primary objective of this study is to assess whether basal cell carcinoma (BCC) lesions surgically treated with curettage, followed by imiquimod 5% cream as postsurgical adjuvant therapy, will have an improved cure rate over the ED/C historical norm of approximately 70% at 1-year posttreatment follow-up. A secondary objective is to assess cosmetic outcome.

DETAILED DESCRIPTION:
This was an open-label, phase IIIb, multicenter, single arm, historical-controlled study. Biopsy-confirmed BCC lesions (1 per subject) were excised by curettage, with no electrodessication. Approximately 1 week later, treatment with imiquimod 5% cream was initiated. Imiquimod was applied to the target BCC once daily, 5 times per week (5x/week) for up to 6 weeks. Rest periods were allowed as needed. Subjects reported to the study center at treatment weeks 1, 2, and 6, and posttreatment at weeks 12, 26, and 52. At treatment week 6 and all posttreatment visits, the investigator clinically assessed the target site for tumor clearance and cosmetic outcome. A template made at initiation and created from clear plastic overlay aided in locating the target tumor site. If the investigator identified a lesion that had occurred or recurred at the target site, the subject was discontinued from the study and counted as a recurrence/persistence (R/P).

ELIGIBILITY:
Inclusion Criteria:

* Basal cell carcinoma

Exclusion Criteria:

* Psoriasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2004-01; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Number of subjects with recurrence | 1 year posttreatment
  Primary variable was the proportion of subjects with recurrence/persistence (R/P)of BCC at 1 year posttreatment

SECONDARY OUTCOMES:
Cosmetic outcome of the target lesion | 1 year posttreatment
  The cosmetic outcome of the target lesion at 1 year posttreatment was the secondary efficacy measurement. The investigator judged cosmetic outcome by using a visual analog scale (VAS) to assess the parameters of hypo- and hyperpigmentation,roughness, scarring, and overall skin health and appearance.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Grass Valley, California
  - Loma Linda, California
  - New York, New York

REFERENCES:
- [Background] Rigel DS, Torres AM, Ely H. Imiquimod 5% cream following curettage without electrodesiccation for basal cell carcinoma: preliminary report. J Drugs Dermatol. 2008 Jan;7(1 Suppl 1):s15-6. PMID 18277458